CLINICAL TRIAL: NCT04524767
Title: Community Partnered Participatory Approach to Implement Depression Screening in Black Churches
Brief Title: Depression Screening in Black Churches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Olajide Williams, Vice Chair of the Department of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AAAT1474; 1R01MH121590-01A1 (NIH)
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT (Experimental): SBIRT will involve screening with the Patient Health Questionnaire-9 (PHQ-9); brief intervention with Motivational Interviewing (MI); and referral to specialty treatment, as needed for subjects with persistent depressive symptoms.
  Interventions: Behavioral: SBIRT
- Referral As Usual (Active Comparator): Referral as Usual will involve distributing depression educational materials (e.g., from the National Institute of Mental Health) and contact information for treatment providers in our target community
  Interventions: Behavioral: Referral as Usual

INTERVENTIONS:
Behavioral: SBIRT — Screening Brief Intervention and Referral to Treatment (SBIRT) is an evidence-based approach designed to provide screening, brief intervention, and referral to more intensive treatment for people at risk of developing mental disorders, including depression. SBIRT is composed of three core components: screening with a validated instrument, brief intervention, referral to treatment. Motivational Interviewing (MI) is the brief intervention most commonly used in SBIRT. MI is an empirically tested, person-centered, behavior change intervention designed to guide, elicit, and strengthen motivation for change. Subjects enrolled in the experimental SBIRT arm will receive up to a maximum of six sessions of MI.
  Arms: SBIRT
Behavioral: Referral as Usual — We will utilize depression educational brochures describing the nine hallmark symptoms of depression symptoms and the importance of seeking treatment from pamphlets from the National Institute of Mental Health (NIMH). Subjects will also receive a list of referral sites in the study's catchment area of Upper Manhattan
  Arms: Referral As Usual

SUMMARY:
The overall aim of this study is to employ Community Health Workers (CHWs) to screen for depression in 30 Black churches and compare the effectiveness of Screening, Brief Intervention, and Referral to Treatment (SBIRT) (Intervention arm) to Referral As Usual (Control arm) on treatment engagement for depression. The investigators will assess patient-level outcomes (Mental-Health Related Quality of Life and depressive symptoms) at 3- and 6-months post-screening and conduct a mixed-methods process evaluation to assess multi-level facilitators and barriers of screening uptake.

DETAILED DESCRIPTION:
African American adults (AAs), compared to White adults, are half as likely to be screened for depression in primary care settings. Disparities in depression screening contribute to poor clinical outcomes, as AAs with depression are more disabled, sicker longer, and less likely to seek treatment compared to Whites. Black churches are trusted settings that provide "de facto" mental health services for depression. Indeed, in the first study of its kind, the study team found that 20% of adults in Black churches screened positive for depression using the Patient Health Questionnaire-9 (PHQ-9). However, no subjects with a positive screen (PHQ-9 ≥10) accepted a treatment referral when offered by research coordinators onsite for each screening.

Community Health Workers (CHWs), who are trusted para-professionals from the target community, may bridge the gap between depression screening and treatment. The investigators have trained and certified 102 CHWs from 42 Black churches in Harlem, New York to deliver an evidence-based intervention called Screening, Brief Intervention, and Referral to Treatment (SBIRT), which is centered on culturally tailored Motivational Interviewing (MI). Thus, the scientific premise of this study is that employing CHWs to implement depression screening in Black churches will bridge the gap between church-based depression-screening and engagement with clinical services.

Using a Hybrid Type 1 Effectiveness-Implementation design, the investigators propose a 2-arm, mixed-methods Cluster-Randomized Controlled Trial within 30 Black churches our CHWs currently attend. Based on our pilot data, the investigators expect 20% of adults (n=600) to have a positive depression screen. Adults will be randomized based on church study site to either SBIRT (n=15 churches) or Referral As Usual (RAU, n=15 churches). The investigators will then compare the effectiveness of SBIRT (Intervention arm) to RAU (Usual Care arm) on treatment engagement (primary outcome), defined as attending a depression-related clinical visit for which the subject reported receiving information, referral, counseling, or medication for depression (Aim 1). The investigators will then compare changes in Mental Health Related Quality of Life and depressive symptoms (secondary outcomes) at 3- and 6-months post-screening (Aim 2). Finally, the investigators will conduct a concurrent, mixed-methods (qualitative-quantitative) process evaluation to assess contextual facilitators and barriers of screening and referral (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Fluent in English
* Patient Health Questionnaire-9 score and/or Generalized Anxiety Disorder-7 ≥ 10

Exclusion Criteria:

* Reporting active suicidality, or verbally endorsing homicidal ideation or psychotic symptoms
* Currently receiving formal mental health treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Treatment Engagement | Measured at 3-months post-screening
  Attendance at a depression-related clinical visit for which the subject reported receiving information, referral, counseling, or medication for depression as assessed by the Community Partners in Care Health Services Use Scale
Treatment Engagement | Measured at 6-months post-screening
  Attendance at a depression-related clinical visit for which the subject reported receiving information, referral, counseling, or medication for depression as assessed by the Community Partners in Care Health Services Use Scale

SECONDARY OUTCOMES:
Change in Depressive Severity | Measured at 3- and 6-months post-screening
  16-Item Quick Inventory of Depressive Symptomatology (QIDS-SR). The QIDS-SR is a validated self-report measure that assesses depressive severity. Scores range from 0 to 27 (worse outcome).
Change in Depressive Symptoms | Measured at 3- and 6-months post-screening
  NIH PROMIS-Depression Scale. This 8-item assessment is a composite of depressive symptoms from the Patient-Reported Outcomes Measurement Information System.
Change in Mental Health-Related Quality of Life | Measured at 3- and 6-months post-screening
  The Mental Health Component Summary Score of the 12-Item Medical Outcomes Study Short-Form (SF-12). The SF-12 is a commonly used measure of functioning, with standardized mean score of 50 and standard deviation of 10.
Change in Anxiety Severity | Measured at 3- and 6-months post-screening
  Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is a self-report measure that assesses anxiety symptoms. Scores range from 0 to 21 (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Olajide Williams, MD, MS, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through submission of study findings to peer-reviewed journals. De-identified data will also be shared at community forums and academic conferences.
Supporting Information: Study Protocol
Time Frame: Data will be available six months after publication in a peer-reviewed journal article.
Access Criteria: The study Co-Primary Investigators, Drs. Sidney Hankerson and Olajide Williams, will create criteria and review requests for data sharing access. Data will be available to analyze waht types of clinical and demographic factors impact study outcomes.

REFERENCES:
- [Background] Hankerson SH, Lee YA, Brawley DK, Braswell K, Wickramaratne PJ, Weissman MM. Screening for Depression in African-American Churches. Am J Prev Med. 2015 Oct;49(4):526-33. doi: 10.1016/j.amepre.2015.03.039. Epub 2015 Jul 29. PMID 26232907
- [Background] Bray JW, Del Boca FK, McRee BG, Hayashi SW, Babor TF. Screening, Brief Intervention and Referral to Treatment (SBIRT): rationale, program overview and cross-site evaluation. Addiction. 2017 Feb;112 Suppl 2:3-11. doi: 10.1111/add.13676. PMID 28074566
- [Background] Boutin-Foster C, Offidani E, Kanna B, Ogedegbe G, Ravenell J, Scott E, Rodriguez A, Ramos R, Michelen W, Gerber LM, Charlson M. Results from the Trial Using Motivational Interviewing, Positive Affect, and Self-Affirmation in African Americans with Hypertension (TRIUMPH). Ethn Dis. 2016 Jan 21;26(1):51-60. doi: 10.18865/ed.26.1.51. PMID 26843796
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Wells KB, Jones L, Chung B, Dixon EL, Tang L, Gilmore J, Sherbourne C, Ngo VK, Ong MK, Stockdale S, Ramos E, Belin TR, Miranda J. Community-partnered cluster-randomized comparative effectiveness trial of community engagement and planning or resources for services to address depression disparities. J Gen Intern Med. 2013 Oct;28(10):1268-78. doi: 10.1007/s11606-013-2484-3. Epub 2013 May 7. PMID 23649787
- [Derived] Hankerson SH, Shelton R, Weissman M, Wells KB, Teresi J, Mallaiah J, Joshua A, Williams O. Study protocol for comparing Screening, Brief Intervention, and Referral to Treatment (SBIRT) to referral as usual for depression in African American churches. Trials. 2022 Jan 31;23(1):93. doi: 10.1186/s13063-021-05767-8. PMID 35101100